CLINICAL TRIAL: NCT04981080
Title: Prevalence of Detrusor Underactivity and Bladder Outlet Obstruction in Women With and Without Symptoms of Voiding Dysfunction
Brief Title: DU and BOO in Women With and Without Symptoms of VD
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202105082RINA
Record Dates: First submitted 2021-07-20; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Detrusor Underactivity; Bladder Outlet Obstruction
Keywords: detrusor underactivity; bladder outlet obstruction; voiding dysfunction
MeSH Terms: conditions — Urinary Bladder, Underactive; Urinary Bladder Neck Obstruction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptom of voiding dysfunction: Women with lower urinary tract symptoms including voiding symptoms but without cystocele who visited the urogynecological department of a medical center for urodynamic evaluation were reviewed
  Interventions: Diagnostic Test: Urodynamic study
- No symptom of voiding dysfunction: Women with lower urinary tract symptoms but without cystocele or voiding symptoms who visited the urogynecological department of a medical center for urodynamic evaluation were reviewed
  Interventions: Diagnostic Test: Urodynamic study

INTERVENTIONS:
Diagnostic Test: Urodynamic study — The urodynamic assessment, including noninstrumented uroflowmetry, filling cystometry with 35°C distilled water at a rate of 60 mL/sec, a pressure flow study, and urethral pressure profilometry, was performed with the patient in a sitting position according to the recommendations by the International Continence Society.

SUMMARY:
Women with symptoms of voiding dysfunction may be associated with detrusor underactivity or bladder outlet obstruction. However, the prevalence of detrusor underactivity and bladder outlet obstruction remained obscure. Thus, the aim of this study was to elucidate the prevalence of detrusor underactivity and bladder outlet obstruction in women with and without symptoms of voiding dysfunction.

DETAILED DESCRIPTION:
Between February 2005 and December 2020, all women with lower urinary tract symptoms but without cystocele who visited the urogynecological department of a medical center for urodynamic evaluation were reviewed. Those women who have no complete data of maximum flow rate, voided volume, post-void residual volume and detrusor pressure at maximum flow rate were excluded from this study. Detrusor underactivity was defined when the detrusor pressure at maximum flow rate was less than 20 cmH2O, the maximum flow rate was less than 15 mL/s, and the bladder voiding efficiency was less than 90 %. Bladder outlet obstruction was defined when the the detrusor pressure at maximum flow rate was not less than 40 cmH2O, and the maximum flow rate was less than 12 mL/s. Those women without detrusor interactivity or bladder outlet obstruction were allocated to the non-DU/BOO group.

STATA software was used for statistical analysis. Chi2 test, univariate and multivariable logistic regression test were used for statistical analysis as appropriate. A p < 0.05 was considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Women with lower urinary tract symptoms
* Complete urodynamic study

Exclusion Criteria:

* Advanced cystocele
* After surgery for cystocele repair
* Chronic infection
* Incomplete data

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with lower urinary tract symptoms but without cystocele who visited the urogynecological department of a medical center for urodynamic evaluation
Sampling Method: Non-Probability Sample
Enrollment: 1886 (Actual)
Dates: Start 2005-02-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Detrusor underactivity | February 2005 and December 2020
  The detrusor pressure when maximal flow rate was less than 20 cmH2O, the maximal flow rate was less than 15 mL/s, and the bladder voiding efficiency was less than 90 %
Bladder outlet obstruction | February 2005 and December 2020
  The detrusor pressure when maximal flow rate was not less than 40 cmH2O, and the maximal flow rate was less than 12 mL/s

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data is available under reasonable request

REFERENCES:
- [Result] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Result] Choi YS, Kim JC, Lee KS, Seo JT, Kim HJ, Yoo TK, Lee JB, Choo MS, Lee JG, Lee JY. Analysis of female voiding dysfunction: a prospective, multi-center study. Int Urol Nephrol. 2013 Aug;45(4):989-94. doi: 10.1007/s11255-013-0475-2. Epub 2013 May 31. PMID 23722818
- [Result] Retraction: Current Concepts in Voiding Dysfunction and Dysfunctional Voiding: A Review from a Urogynaecologist's Perspective. J Midlife Health. 2018 Jan-Mar;9(1):50. doi: 10.4103/0976-7800.227258. PMID 29628732
- [Result] Robinson D, Staskin D, Laterza RM, Koelbl H. Defining female voiding dysfunction: ICI-RS 2011. Neurourol Urodyn. 2012 Mar;31(3):313-6. doi: 10.1002/nau.22213. Epub 2012 Mar 13. PMID 22415792
- [Result] Hsiao SM, Lin HH, Kuo HC. Videourodynamic Studies of Women with Voiding Dysfunction. Sci Rep. 2017 Jul 28;7(1):6845. doi: 10.1038/s41598-017-07163-2. PMID 28754926
- [Result] Lukacz ES, DuHamel E, Menefee SA, Luber KM. Elevated postvoid residual in women with pelvic floor disorders: prevalence and associated risk factors. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Apr;18(4):397-400. doi: 10.1007/s00192-006-0164-0. Epub 2006 Jun 28. PMID 16804634
- [Result] Milleman M, Langenstroer P, Guralnick ML. Post-void residual urine volume in women with overactive bladder symptoms. J Urol. 2004 Nov;172(5 Pt 1):1911-4. doi: 10.1097/01.ju.0000140502.34334.75. PMID 15540753